CLINICAL TRIAL: NCT01753596
Title: Assessment of Tear Film Thickness by Optical Coherence Tomography in Healthy Subjects and Subjects With Dry Eye Disease
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: OPHT-200612
Record Dates: First submitted 2012-12-07; First posted 2012-12-20 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Dry Eye Syndrome
Keywords: topical lubricants; tear film thickness; break up time; ocular surface disease index; Schirmer I test
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 30 healthy subjects (Experimental): Subjects will receive 1 drop of Genteal HA eye drops in one randomly chosen eye, the other eye will receive placebo
  Interventions: Device: GENTEAL HA® Eye Drops (NOVARTIS, Switzerland); Other: Physiological Sodium Chloride solution (0,9%)
- 30 patients with dry eye syndrome (Experimental): Patients will receive 1 drop of Genteal HA eye drops in one randomly chosen eye, the other eye will receive placebo
  Interventions: Device: GENTEAL HA® Eye Drops (NOVARTIS, Switzerland); Other: Physiological Sodium Chloride solution (0,9%)

INTERVENTIONS:
Device: GENTEAL HA® Eye Drops (NOVARTIS, Switzerland)
Other: Physiological Sodium Chloride solution (0,9%) — Placebo

SUMMARY:
Dry eye syndrome (DES) is a highly prevalent ocular condition with severe consequences for the patients reaching from ocular discomfort in its simplest form up to visual impairment and corneal ulceration in severe cases. Data from epidemiological studies indicate that DES is a common disease, especially in the elderly population, affecting up to 20% of adults aged 45 years or older. Topical lubricants are a mainstay of therapy, but data on its effect on tear film thickness and the corneal residence time are lacking.

Recently, a new objective method for assessment of tear film thickness by optical coherence tomography has been developed. The present study aims to investigate the corneal residence time of an established topical lubricant compared to placebo in patients with DES and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for healthy subjects:

* Men and women aged over 18 years
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 6 Dpt
* Schirmer I test > 10 mm and BUT > 10 sec

Inclusion criteria for patients with dry eye syndrome:

* Men and women aged over 18 years
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant except DES
* Normal ophthalmic findings, ametropia < 6 Dpt
* History of dry eye syndrome for at least 3 months
* Tear Break Up Time (BUT) < 10 seconds or Schirmer I test < 7 mm
* At least 2 symptoms of dry eye syndrome (foreign body sensation, burning, photophobia, blurred vision, pain, itching)
* Normal ophthalmic findings except dry eye syndrome

Exclusion Criteria:

* Regular use of medication (except contraceptives), abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Ametropia >= 6 Dpt
* Pregnancy
* Difference of more than 3 mm in Schirmer I test or difference of > 3 sec in BUT between the two eyes
* Known medical history of allergy, hypersensitivity or poor tolerance to any components of the medication or medical product used in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Tear film thickness | change from baseline to 1 hour after administration

SECONDARY OUTCOMES:
Schirmer I Test | 1 day
  once on the study day
Tear Break Up Time | 1 day
  once on the study day
Ocular Surface Disease Index | 1 day
  once on the study day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Vienna, Austria